CLINICAL TRIAL: NCT02166658
Title: A Phase II Study of Cabazitaxel for Patients With Breast or Lung Cancer and Recurrent or Progressive Brain Metastases - Cabazitaxel for Brain Metastases (CaBaMet)
Brief Title: A Study of Cabazitaxel for Patients With Breast or Lung Cancer and Recurrent or Progressive Brain Metastases - Cabazitaxel for Brain Metastases (CaBaMet)
Acronym: CaBaMet
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After a recruitment of more than 2 years, only 8 patients have been registered.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: ClinAssess GmbH (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-ZNS-0113; 2013-005545-37 (EudraCT Number); CABAZL06457 (Other: Sanofi-Aventis)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer; Lung Cancer; Recurrent Brain Metastases; Progressive Brain Metastases
Keywords: Patients with breast or lung cancer and recurrent or progressive brain; metastases
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Brain Neoplasms; Recurrence; Neoplasm Metastasis | interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Patients receive Cabazitaxel 25 mg/m2 i.v. infusion. This trial is a single arm trial.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel 25 mg/m2 i.v. infusion (infusion time about 1h) on D1 of each 21-day cycle. Continuation of treatment until progression of brain metastases or unacceptable toxicity.
  Other Names: XRP6258, RPR116258A

SUMMARY:
Patients suffering from histologically or cytologically confirmed stage IV lung or breast cancer with progressive or recurrent brain metastases after prior external beam radiotherapy will receive treatment with cabazitaxel until progression of brain metastases (BM) or unacceptable toxicity.

DETAILED DESCRIPTION:
Cabazitaxel is a new taxane compound that exhibited a broad spectrum of in vivo antitumor activity, not only in docetaxel - sensitive tumor models, but also in tumors models in which docetaxel was poorly or not active. In contrast to other taxanes, cabazitaxel has the ability to cross the blood-brain-barrier. Marked antitumor activity was obtained in nude mice bearing intracranial glioblastomas. Consequently, there is a good rationale to investigate cabazitaxel in patients with breast or lung cancer and recurrent or progressive brain metastases.

The primary object of the study is to measure objective tumor response of brain metastases for patients with breast or lung cancer and recurrent or progressive brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years of age)
2. Histologically or cytologically confirmed stage IV lung or breast cancer with progressive or recurrent brain metastases
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Prior external beam radiotherapy (WBRT or SRS) of BM Patients suffering from small cell lung cancer (SCLC) who have been treated with chemotherapy and prophylactic cranial radiotherapy may be also enrolled.
5. At least one two-dimensional measurable lesion on brain MRI
6. Life expectancy at least 3 months
7. Females of childbearing potential (FCBP) must have a negative pregnancy test within 7 days of the first application of study treatment and must agree to use effective contraceptive birth control measures (Pearl Index < 1) during the course of the Trial. A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 year, or unless she is surgically sterile.
8. Males must agree to use effective contraception (Pearl Index < 1) during the course of the trial and for at least 6 months after last administration of study medication cabazitaxel. In addition males must agree to prevent contact with the ejaculate by another person throughout study treatment.

Exclusion Criteria:

1. Prior chemotherapy or targeted therapy (e.g. erlotinib, bevacizumab) for brain metastases
2. Any chemotherapy or targeted tumor therapy within two weeks of study inclusion or concomitantly
3. Any antihormonal tumor treatment within two weeks of study inclusion or concomitantly
4. Time interval to prior external beam radiotherapy less than 2 weeks
5. Suspected or known leptomeningeal disease
6. Peripheral neuropathy ≥ grade 2
7. Inadequate organ and bone marrow function as evidenced by:

   * Absolute neutrophil count (ANC) < 1.5 x 10*9/L;
   * Hemoglobin < 10.0 g/dL;
   * Platelet count < 100 x 10*9/L;
   * Total bilirubin ≥ 1 x upper limit of normal (ULN);
   * AST/GOT and/or ALT/GPT ≥ 1.5 x ULN;
   * Serum creatinine > 1.5 x ULN. If creatinine 1.0 - 1.5 x ULN; creatinine clearance has to be calculated according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula and patients with creatinine clearance < 60 mL/min must be excluded
8. Other inadequate organ function according to investigator's discretion
9. History of hypersensitivity reaction to docetaxel
10. History of hypersensitivity reaction to polysorbate 80 containing drugs
11. Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
12. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week washout period is necessary for patients who are already on these treatments; see also Section 10 and Appendix 3 and 4; dexamethasone is allowed)
13. Recently received or planned vaccination against yellow fever during study treatment
14. Pregnant or breast feeding females
15. Participation in any other clinical trial or treatment with any experimental drug within 28 day before enrolment to the study or during study participation until the end of treatment visit
16. Previous or concurrent tumor other than underlying tumor disease (breast or lung cancer) with the exception of cervical cancer in situ, adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, superficial bladder tumors (Ta,Tis, and T1) or any curatively treated tumors > 5 years prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Objective tumor response of brain metastases | approx. 12 month
  Objective tumor response of brain metastases (Complete response (CR) or partial response (PR) or at least a minor response (MR; 25-50% reduction) according to WHO criteria1,2 and Iwamoto3 confirmed by magnetic resonance imaging (MRI))

SECONDARY OUTCOMES:
Overall Survival | approx. 12 month
  Efficacy measure
Progression free-survival for brain metastases | approx. 12 month
  Efficacy measure
progression-free survival for extracerebral tumor disease | approx. 12 month
  Efficacy measure
Time to treatment failure of brain metastases | 12 month
  Efficacy measure
Quality of life | approx. 12 month
  Efficacy measure, assessed with EORTC QLQ-C30 and additional module BN20 questionnaire
Type, incidence and severity of adverse events | approx. 12 month
  Safety measure
Dose reduction or discontinuation of study drug cabazitaxel due to adverse events | approx. 12 month
  Safety measure

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kullmann, Prof. Dr., Principal Investigator — Kliniken Nordoberpfalz AG, Klinikum Weiden, Medizinische Kliniken I
Locations (1):
- Kliniken Nordoberpfalz, AG Klinikum Weiden, Medizinische Kliniken I, Weiden, Bavaria, Germany

REFERENCES:
- See also: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de